CLINICAL TRIAL: NCT04571502
Title: Integration of Health Information Technology and Promotion of Personhood in Family-Centered Dementia Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01AG068572 (NIH); NIH Award R01AG068572 (Other Grant/Funding Number: NIA)
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Neurocognitive Disorders; Alzheimer Disease; Caregiver
Keywords: Health technology; Assistive and Alternative Communication Device; Family Centered Care; Personhood
MeSH Terms: conditions — Neurocognitive Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors will not be involved with the intervention implementation and study participants will be asked not to reveal their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Intervention (Experimental): Dyads (caregiver, PWD) randomly assigned to the experimental arm will have access to the newly developed My PATI app. Providers' will receive information via the app.
  Interventions: Other: My PATI ( Person Assisted Touchscreen Interface)
- Usual Care (No Intervention): Dyads (caregiver, PWD) randomly assigned to the usual care condition will receive usual care from the memory clinic.

INTERVENTIONS:
Other: My PATI ( Person Assisted Touchscreen Interface) — My PATI was designed to support communication between PWD and their caregiver, and healthcare provide; promotes person centered care by giving the PWD their voice and specifically by supporting the PWD in expressing their experiences , needs, preferences in care activities (e.g., food choices, clothing), and entertainment ( personalized pictures, videos , and music). My PATI has multiple features including allowing the caregiver to assess symptoms of the PWD using clinical assessments, which can be shared with the healthcare provider. The clinical trial evaluates the impact of the My PATI interface that relies on touchscreen technology ( two interfaces one for PWD that can be used independently or with assistance, and a 2nd caregiver interface for customization ). The comparison group will receive usual care.
  Arms: Full Intervention

SUMMARY:
Alzheimer's disease and related dementias (ADRD) are leading causes of disability and often result in communication deficits of the person with dementia (PWD) that can complicate ADRD caregiving and clinical care. The research team will work with stakeholders to develop and design a personalized Assistive and Alternative Communication (AAC) device that relies on information technology (IT) and touchscreens to promote communication and personhood for PWD about their care preferences and experiences. This study will integrate the AAC into an existing health IT intervention that already facilitates clinical communication between caregivers and providers of PWD. A clinical trial will be conducted to evaluate outcomes of 58 dyads (PWD/caregivers) and their health care provider utilizing the My PATI (My Person Assisted Touchscreen Interface)intervention as an adjunct to care and care giving for 6 months.

DETAILED DESCRIPTION:
The target enrollment for the clinical trial is 58 dyads of caregivers and people with dementia (PWD), where 58 unique dyads of caregivers/PWD will participate. The team plans to enroll a total of 58 dyads across two participating clinical sites. Participants will be randomly assigned to either the full intervention or a control condition for a period of 6 months, where they will be asked to communicate clinical and other relevant information with one another as part of regular caregiving and clinical care activities. Several psychosocial outcome variables for providers, caregivers, and PWD will be assessed. We will compare outcomes based on group assignment and different amounts and patterns of use of the MyPATI (e.g., minimal/non-users versus frequent users). The primary outcome variables are quality of life for caregivers and PWD. The research team will recruit an estimated 15 healthcare providers across both sites at the end of study to assess their experience with My PATI using open and closed ended queries.

ELIGIBILITY:
Inclusion Criteria

Caregivers:

* Regular access to the internet (via computer or smartphone) and telephone
* 21 years-old or older
* Providing caregiving activities (Activities of Daily Living and/or Instrumental Activities of Daily Living) for an average of 2 hours or more per day of direct assistance or supervision for a person with ADRD
* Speak and understand English or Spanish.

Care Recipient:

* 60 years or older
* Speak and understand English or Spanish
* Have an established diagnosis of a Neurocognitive Disorder (Alzheimer's disease, vascular dementia, frontotemporal dementia, Lewy body dementia or Parkinson's disease dementia)
* Receive a score on the Mini Mental Status Exam of less than 24
* Be able to complete the eligibility vision screen.

Healthcare Providers:

* Provide ongoing healthcare and support services to PWD and their families.

Exclusion Criteria

Caregivers:

* Provide care to a PWD living in an assisted living facility or nursing home
* Plan for the PWD to be placed in a long-term care facility during the study period
* Plan to end their role as caregiver within 6 months of study enrollment
* Have their own major medical conditions affecting independent functioning (e.g. illness or disability) or cognitive impairment
* Do not speak and read English or Spanish
* Have known active suicidal ideation

Care Recipients:

* Significant visual or hearing impairment (with supports)
* Known active suicidal ideation
* Schizophrenia diagnosis

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life In Alzheimer's disease- Care Recipient and Caregiver (proxy-interview) | Baseline, 3-months, 6- months
  The 13-item QOL-AD scale uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the care recipient's physical health, mood, relationships, activities, and ability to complete tasks. The Care Recipient (self-assesses) and caregiver (proxy-interview) complete the QOL-AD.
Change in Perceived Change Index- Caregiver QOL | Baseline, 3-months, 6- months
  A 13-item scale that measures caregiver appraisals of self-improvement or decline in distinct areas of well- being. Caregiver indicates whether each item has become worse, stayed the same, or improved in the past month: feeling rested, ability to have time for yourself, and feelings of being upset. The total and subscales (Affect, Somatic, and Ability to Manage)

SECONDARY OUTCOMES:
Change in PATIENT HEALTH QUESTIONNAIRE (PHQ-9)- Caregiver | Baseline, 3-months, 6- months
  The 9-item Patient Health Questionnaire (PHQ-9) includes nine items that correspond to each of the nine symptoms of major depression from the Diagnostic and Statistical Manual of Mental Disorders. The PHQ-9 scores range from 0 to 27 (increasing score correlates with increasing depression severity) and each of the 9 items is scored from 0 to 3, indicating "how often a symptom is bothersome."
Change in The Positive Aspects of Caregiving Scale- Caregiver | Baseline, 3-months, 6- months
  The Positive Aspects of Caregiving Scale (Tarlow et al., 2004) assesses positive feelings resulting from care provision among family caregivers of older adults with functional limitations. Each of the 9 items on the scale asks about potential benefits from caregiving for the caregivers.
Change in Zarit Caregiver Burden Inventory-22 items (ZBI-22)- Caregiver | Baseline, 3-months, 6-months
  The ZBI-22 (22 items) assesses common stressors experienced by dementia caregivers. A list of statements which reflect how people sometimes feel when taking care of another person are presented and caregivers are queried about how often they felt that way (never, rarely, sometimes, quite frequently, or nearly always).
Change in 12 Item Short-Form Health Survey (SF-12) - Caregiver | Baseline,6-months
  The SF-12 is a validated, shortened version of the The RAND Health Care 36-Item Health Survey that includes 7 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
Change in The Revised Memory and Behavior Problems Checklist - Caregiver interviewed about Care Recipient | Baseline, 6-months
  The Revised Memory and Behavior Problems Checklist, a 24-item caregiver-reported measure of observable memory difficulties and behavior problems in patients along with a parallel assessment of the caregiver's reaction to these behavioral problems. The checklist is a reliable and valid assessment that asks the caregiver to rate the frequency of care recipient problems (0 = never occurred to 4 = daily or more often) within three subscales (i.e., memory-related, depression, and disruptive behaviors). The caregiver rates the frequency of each behavior problem during the past week and his/her reaction to the behavior (i.e., how bothered or upset the caregiver feels when the behavior occurs [0 = not at all to 4 = extremely bothered]).
Change in Oberved PHQ-9 Caregiver Interviewed about Care Recipient | Baseline, 6-months
  The PHQ-9 observed version is a depression severity measure used for screening for mood disorders in nursing home populations (Saliba et al, 2012). The 9 signs and symptoms are assessed by interviewing an informant about their observations of client symptoms over the previous 2 weeks.
Change in Geriatric Depression Scale (GDS-15)- Care Recipient | Baseline, 6-months
  The 15-item Geriatric Depression Scale (GDS-15) is a depression screening tool developed for use in older adults. It had been validated for community-dwelling, hospitalized, and institutionalized older adults. The GDS-15 has a yes-no format. Scores range from 0 to 15; the higher the score the more likely the individual is experiencing depression.
Change in Partner-Patient Questionnaire for Shared Activities-Caregiver interviewed about relationship with Care Recipient | Baseline, 3 Months, 6 Months
  The PPQSA was constructed to measure the extent to which the AD patient's mood and mental state interfered with the patient-partner relationship.
Change in Functional Linguistic Communication Inventory (FLCI)- Care Recipient | Baseline
  Functional Linguistic Communication Inventory (FLCI) is a standardized instrument for evaluating functional communication in persons with moderate and severe dementia. A number of domains assessed included: Greeting and naming, Answering questions, Writing, Sign comprehension, Object-to-picture matching, Word reading and comprehension, Reminiscing, Following commands, Pantomime, Gesture, and Conversation.
My PATI Usage - Links clicked on the app, resources accessed | 6 months
  The research team will track user actions ( provider, caregiver, care recipient) on the Web and Android/iphone operating system Apps, such as login, logout, viewing of educational material, taking a health assessment, or contacting the provider.
Provider Interviews | 6 months
  The research team will conduct interviews with the providers who are participating with intervention dyads. The interview questions will include newly-created closed-ended questions, and open-ended qualitative questions that will assess their perceptions of integrating My PATI into clinical workflow (e.g. acceptability of technology, problems experienced, observed benefits); and how use of My PATI influenced clinical/shared decision making and clinical care.
My PATI Usage- Links clicked on the app, resources accessed | 6 months
  The research team will track user actions ( provider, caregiver, care recipient) on the Web and Android/IOS Apps, such as login, logout, viewing of educational material, taking a health assessment, or contacting the provider.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UAB Alzheimer's Risk Assessment and Intervention Clinic, Birmingham, Alabama
  - Miami Jewish Health, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Tarlow BJ, Wisniewskil SR, Belle SH., et al. Positive Aspects of Caregiving: Contributions of the REACH Project to the Development of New Measures for Alzheimer's Caregiving. 2004; 26(4):429-53.
- [Background] Roth DL, Burgio LD, Gitlin LN, Gallagher-Thompson D, Coon DW, Belle SH, Stevens AB, Burns R. Psychometric analysis of the Revised Memory and Behavior Problems Checklist: factor structure of occurrence and reaction ratings. Psychol Aging. 2003 Dec;18(4):906-15. doi: 10.1037/0882-7974.18.4.906. PMID 14692875
- [Background] Brown EL, Ruggiano N, Page TF, Roberts L, Hristidis V, Whiteman KL, Castro J. CareHeroes Web and Android Apps for Dementia Caregivers: A Feasibility Study. Res Gerontol Nurs. 2016 Jul-Aug;9(4):193-203. doi: 10.3928/19404921-20160229-02. Epub 2016 Mar 4. PMID 29977440
- [Background] Brown EL, Agronin ME, Stein JR. Interventions to Enhance Empathy and Person-Centered Care for Individuals With Dementia: A Systematic Review. Res Gerontol Nurs. 2020 May 1;13(3):158-168. doi: 10.3928/19404921-20191028-01. Epub 2019 Nov 11. PMID 31697393
- [Background] Ruggiano N, Brown EL, Li J, Scaccianoce M. Rural Dementia Caregivers and Technology: What Is the Evidence? Res Gerontol Nurs. 2018 Jul 1;11(4):216-224. doi: 10.3928/19404921-20180628-04. PMID 30036405
- [Background] Brown EL, Ruggiano N, Li J, Clarke PJ, Kay ES, Hristidis V. Smartphone-Based Health Technologies for Dementia Care: Opportunities, Challenges, and Current Practices. J Appl Gerontol. 2019 Jan;38(1):73-91. doi: 10.1177/0733464817723088. Epub 2017 Aug 4. PMID 28774215
- [Background] Ruggiano N, Brown EL, Shaw S, Geldmacher D, Clarke P, Hristidis V, Bertram J. The Potential of Information Technology to Navigate Caregiving Systems: Perspectives from Dementia Caregivers. J Gerontol Soc Work. 2019 May-Jun;62(4):432-450. doi: 10.1080/01634372.2018.1546786. Epub 2018 Nov 13. PMID 30422754
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Teri L, Truax P, Logsdon R, Uomoto J, Zarit S, Vitaliano PP. Assessment of behavioral problems in dementia: the revised memory and behavior problems checklist. Psychol Aging. 1992 Dec;7(4):622-31. doi: 10.1037//0882-7974.7.4.622. PMID 1466831
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Bayles KA, Tomoeda CK. FLCI: Functional Linguistic Communication Inventory. Canyonlands Publishing, Incorporated; 1994.
- [Derived] Brown EL, Ruggiano N, Roberts L, Clarke PJ, Davis DL, Agronin M, Geldmacher DS, Hough MS, Munoz MTH, Framil CV, Yang X. Integration of Health Information Technology and Promotion of Personhood in Family-Centered Dementia Care: Intervention Trial. Res Gerontol Nurs. 2021 Sep-Oct;14(5):225-234. doi: 10.3928/19404921-20210825-02. Epub 2021 Sep 1. PMID 34542347